CLINICAL TRIAL: NCT06259578
Title: Immunobridging Study: Immunogenicity and Safety of INAVAC (Vaksin Merah Putih - UNAIR SARS-CoV-2 (Vero Cell Inactivated)) Vaccine as Homologue Booster in Adult Subjects in Indonesia
Brief Title: UNAIR Inactivated COVID-19 Vaccine as Homologue Booster (Immunobridging Study)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Universitas Airlangga (Other); Bioxis Pharmaceuticalls (Industry); Indonesia-MoH (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNAIR-MP-INAKTIF-BO-009
Record Dates: First submitted 2024-02-05; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Pandemic; COVID-19 Vaccines; COVID-19 Virus Disease
Keywords: Inactivated COVID-19 Vaccine; Immunogenicity; Safety; COVID-19; Indonesia; Immunobridging study; Booster; INAVAC
MeSH Terms: conditions — COVID-19 | interventions — vaksin merah putih - UA SARS-CoV-2 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INAVAC (Vaksin Merah Putih - UA-SARS CoV-2 (Vero Cell Inactivated) 5 μg (Experimental): The study product is provided in the form of liquid in vial single dose (0.5 ml). The vaccine will be given 1 dose (0.5 ml) once.
  Interventions: Biological: INAVAC (Vaksin Merah Putih - UA- SARS CoV-2 (Vero Cell Inactivated) 5 μg

INTERVENTIONS:
Biological: INAVAC (Vaksin Merah Putih - UA- SARS CoV-2 (Vero Cell Inactivated) 5 μg — 1 dose of 0.5 ml containing inactivated SARS-CoV-2 virus (5 μg ), Tween 80, histidine, Polysorbate 80, Aluminium hydroxide gel, and sodium chloride

SUMMARY:
The goal of this open-label clinical trial is to evaluate the safety and immunogenicity of INAVAC (Vaksin Merah Putih - UNAIR SARS-CoV-2 (Vero Cell Inactivated)) Vaccine as Homologue Booster in Adult Subjects in Indonesia. The main question it aims to answer is: "To evaluate the humoral immunogenicity profile at 28 days following vaccination with INAVAC vaccine as homolog booster administered intramuscularly in healthy adults age 18 years and above". Participants will be administered one dose of vaccination for the third dose (booster vaccination) intramuscularly.

DETAILED DESCRIPTION:
This is an open-label trial. There will be only one group in the study. This group will receive the INAVAC vaccine as a booster. The inclusion and exclusion criteria for the subjects are listed below. All subjects will be followed for 6 months. The vaccine will be administered intramuscularly. This study will have one interim and one full analysis report. A Data Safety Monitoring Board will be commissioned for this study to evaluate safety data over the study period and to review any events that meet a specific study pausing rule or any other safety issue that may arise. They will review the 7 and 28-day safety data following the vaccine, and then the 3 and 6-month safety data. The immunogenicity data will be evaluated for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults and elderly, males and females, 18 years of age and above. Healthy status will be determined by the investigator based on medical history, clinical laboratory results, vital sign measurements, and physical examination at screening.
2. Subjects already received 2 (two) doses of INAVAC vaccines (5 ug), mostly during the phase I/II/III clinical trial of this vaccine. The interval between the second primary injection and the booster is 12-18 months.
3. Subjects have been informed properly regarding the study and signed the informed consent form
4. Subjects will commit to comply with the instructions of the investigator and the schedule of the trial
5. Female subjects of childbearing potential must agree to postpone pregnancy from at least 21 days before enrollment and through 6 months after the vaccination.
6. Participants agree not to donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the vaccine.
7. Participants must be willing to provide verifiable identification, have means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another vaccine trial
2. Evolving mild, moderate, and severe illness, especially infectious diseases or fever (axillary temperature 37.5oC or more) concurrently or within 7 days before study vaccination. This includes respiratory or constitutional symptoms consistent with SARS-CoV-2 (cough, sore throat, difficulty in breathing, etc)
3. Known history of allergy to any component of the vaccines
4. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
5. Any autoimmune or immunodeficiency disease/condition
6. Subjects who have received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulin, blood-derived products, long-term corticosteroid - more than 2 weeks, and so on), OR anticipation of the need for immunosuppressive treatment within 6 months after last vaccination. The use of topical or nasal steroids will be permitted. Inhaled glucocorticoids are prohibited.
7. Unstable chronic disease, inclusive of uncontrolled hypertension, congestive heart failure, chronic obstructive pulmonary disease, asthma, chronic urticaria, and diabetes requiring the use of medicine. The final decision regarding this condition will be made by the attending field clinicians or investigators.
8. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives
9. Individuals who previously received any vaccines against Covid-19, other than INAVAC.
10. Subjects already immunized with any other vaccines within 4 weeks prior and expect to receive other vaccines within 60 days following the booster dose
11. Individuals who have a previously ascertained COVID-19 in 1 month (for mild, moderate, or asymptomatic people) or 3 months (for severe COVID-19) before the first recruit of this study, or in close contact in the last 14 days with a confirmed case of Covid-19.
12. Positive test for SARS-CoV-2 (Antigen or PCR) at screening before the vaccination. Testing may be repeated during the screening period if exposure to a positive confirmed case of SARS-CoV-2 is suspected, at the discretion of the investigator.
13. History of alcohol or substance abuse
14. HIV patients.
15. Malignancy patients within 3 years before study vaccination.
16. Any neurological disease or history of significant neurological disorder such as meningitis, encephalitis, Guillain-Barre Syndrome, multiple sclerosis, etc
17. Vital sign abnormalities and clinical laboratory abnormalities as decided by the investigators. Vital sign measurements and clinical laboratory testing may be repeated before the final decision.
18. Women who are pregnant or who plan to become pregnant during the study.
19. Participant has a major psychiatric problem or illness
20. Participant cannot communicate reliably with the investigator
21. Participant has contraindications to intramuscular injection and blood draws, such as bleeding disorders or phobia.
22. The participant had major surgery within 12 weeks before vaccination which will not be fully recovered, or has major surgery planned during the time the participant is expected to participate in the study or within 6 months after the last dose of study vaccine administration.
23. Any condition that in the opinion of the investigators would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine or interpretation of the study results
24. Study team members.
25. Subject planning to move from the study area before the end of the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-08-29 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
Humoral Immune Reponse | 28 days following vaccination
  1. SARS-CoV-2 Neutralization: SARS-CoV-2 neutralizing titers in serum measured by a virus neutralization assay, at 28 days following vaccination with INAVAC vaccine as homologue booster administered intramuscularly in healthy adults age 18 year and above
  2. IgG RBD SARS-CoV-2 antibodies measured by CLIA: analysis of antibodies binding to the SARS-CoV-2 S-protein, at 28 days following vaccination with INAVAC vaccine as homologue booster administered intramuscularly in healthy adults age 18 year and above

SECONDARY OUTCOMES:
Incidence of Adverse Events | 7 days, 28 days, 3 months and 6 months following vaccination
  1. Solicited - clinical (local and systemic) adverse events for 7 and 28 days, 3 and 6 month following vaccination with INAVAC vaccine as homologue booster administered intramuscularly in healthy adults age 18 year and above
  2. Unsolicited adverse events for 7 and 28 days, 3 and 6 months following vaccination with INAVAC vaccine as homologue booster administered intramuscularly in healthy adults age 18 year and above
  3. Serious adverse event (SAE) throughout the study
Humoral Immune Reponse | 3 and 6 months following vaccination
  1. SARS-CoV-2 Neutralization: SARS-CoV-2 neutralizing titers in serum measured by a virus neutralization assay, for 3 and 6 months following vaccination with INAVAC vaccine as homolog booster administered intramuscularly in healthy adults age 18 years and above
  2. IgG RBD SARS-CoV-2 antibodies measured by CLIA: analysis of antibodies binding to the SARS-CoV-2 S-protein, for 3 and 6 months following vaccination with INAVAC vaccine as homolog booster administered intramuscularly in healthy adults age 18 years and above
Exploratory Endpoints | Through study completion, an average of 6 months after the study product administration
  Whole genome sequencing (WGS) of S protein of SARS-CoV-2 virus from positive Covid-19 cases during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Wang Z, Wang G, Lau JY, Zhang K, Li W. COVID-19 in early 2021: current status and looking forward. Signal Transduct Target Ther. 2021 Mar 8;6(1):114. doi: 10.1038/s41392-021-00527-1. PMID 33686059
- [Background] Noh JY, Song JY, Yoon JG, Seong H, Cheong HJ, Kim WJ. Safe hospital preparedness in the era of COVID-19: The Swiss cheese model. Int J Infect Dis. 2020 Sep;98:294-296. doi: 10.1016/j.ijid.2020.06.094. Epub 2020 Jun 30. PMID 32619759
- [Background] Irwin A. What it will take to vaccinate the world against COVID-19. Nature. 2021 Apr;592(7853):176-178. doi: 10.1038/d41586-021-00727-3. No abstract available. PMID 33767468
- [Background] So AD, Woo J. Reserving coronavirus disease 2019 vaccines for global access: cross sectional analysis. BMJ. 2020 Dec 15;371:m4750. doi: 10.1136/bmj.m4750. PMID 33323376
- [Background] Biswas M, Rahaman S, Biswas TK, Haque Z, Ibrahim B. Association of Sex, Age, and Comorbidities with Mortality in COVID-19 Patients: A Systematic Review and Meta-Analysis. Intervirology. 2020 Dec 9:1-12. doi: 10.1159/000512592. Online ahead of print. PMID 33296901
- [Background] Cirrincione L, Plescia F, Ledda C, Rapisarda V, Martorana D, Moldovan RE, Theodoridou K, Cannizzaro E. COVID-19 Pandemic: Prevention and Protection Measures to Be Adopted at the Workplace. Sustainability 2020; 12: 3603
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Background] Palacios R, Patino EG, de Oliveira Piorelli R, Conde MTRP, Batista AP, Zeng G, Xin Q, Kallas EG, Flores J, Ockenhouse CF, Gast C. Double-Blind, Randomized, Placebo-Controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of treating Healthcare Professionals with the Adsorbed COVID-19 (Inactivated) Vaccine Manufactured by Sinovac - PROFISCOV: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Oct 15;21(1):853. doi: 10.1186/s13063-020-04775-4. PMID 33059771
- [Background] Tanriover MD, Doganay HL, Akova M, Guner HR, Azap A, Akhan S, Kose S, Erdinc FS, Akalin EH, Tabak OF, Pullukcu H, Batum O, Simsek Yavuz S, Turhan O, Yildirmak MT, Koksal I, Tasova Y, Korten V, Yilmaz G, Celen MK, Altin S, Celik I, Bayindir Y, Karaoglan I, Yilmaz A, Ozkul A, Gur H, Unal S; CoronaVac Study Group. Efficacy and safety of an inactivated whole-virion SARS-CoV-2 vaccine (CoronaVac): interim results of a double-blind, randomised, placebo-controlled, phase 3 trial in Turkey. Lancet. 2021 Jul 17;398(10296):213-222. doi: 10.1016/S0140-6736(21)01429-X. Epub 2021 Jul 8. PMID 34246358
- [Background] Al Kaabi N, Zhang Y, Xia S, Yang Y, Al Qahtani MM, Abdulrazzaq N, Al Nusair M, Hassany M, Jawad JS, Abdalla J, Hussein SE, Al Mazrouei SK, Al Karam M, Li X, Yang X, Wang W, Lai B, Chen W, Huang S, Wang Q, Yang T, Liu Y, Ma R, Hussain ZM, Khan T, Saifuddin Fasihuddin M, You W, Xie Z, Zhao Y, Jiang Z, Zhao G, Zhang Y, Mahmoud S, ElTantawy I, Xiao P, Koshy A, Zaher WA, Wang H, Duan K, Pan A, Yang X. Effect of 2 Inactivated SARS-CoV-2 Vaccines on Symptomatic COVID-19 Infection in Adults: A Randomized Clinical Trial. JAMA. 2021 Jul 6;326(1):35-45. doi: 10.1001/jama.2021.8565. PMID 34037666
- [Background] Kyriakidis NC, Lopez-Cortes A, Gonzalez EV, Grimaldos AB, Prado EO. SARS-CoV-2 vaccines strategies: a comprehensive review of phase 3 candidates. NPJ Vaccines. 2021 Feb 22;6(1):28. doi: 10.1038/s41541-021-00292-w. PMID 33619260
- [Background] Mendonca SA, Lorincz R, Boucher P, Curiel DT. Adenoviral vector vaccine platforms in the SARS-CoV-2 pandemic. NPJ Vaccines. 2021 Aug 5;6(1):97. doi: 10.1038/s41541-021-00356-x. PMID 34354082
- [Background] Yadav T, Srivastava N, Mishra G, Dhama K, Kumar S, Puri B, Saxena SK. Recombinant vaccines for COVID-19. Hum Vaccin Immunother. 2020 Dec 1;16(12):2905-2912. doi: 10.1080/21645515.2020.1820808. Epub 2020 Nov 24. PMID 33232211
- [Background] Pollard AJ, Bijker EM. A guide to vaccinology: from basic principles to new developments. Nat Rev Immunol. 2021 Feb;21(2):83-100. doi: 10.1038/s41577-020-00479-7. Epub 2020 Dec 22. PMID 33353987
- [Background] Excler JL, Saville M, Berkley S, Kim JH. Vaccine development for emerging infectious diseases. Nat Med. 2021 Apr;27(4):591-600. doi: 10.1038/s41591-021-01301-0. Epub 2021 Apr 12. PMID 33846611
- [Background] Bhattacharya S, Dasgupta R. Smallpox and polio eradication in India: comparative histories and lessons for contemporary policy. Cien Saude Colet. 2011 Feb;16(2):433-44. doi: 10.1590/s1413-81232011000200007. PMID 21340319
- [Background] Jayk Bernal A, Gomes da Silva MM, Musungaie DB, Kovalchuk E, Gonzalez A, Delos Reyes V, Martin-Quiros A, Caraco Y, Williams-Diaz A, Brown ML, Du J, Pedley A, Assaid C, Strizki J, Grobler JA, Shamsuddin HH, Tipping R, Wan H, Paschke A, Butterton JR, Johnson MG, De Anda C; MOVe-OUT Study Group. Molnupiravir for Oral Treatment of Covid-19 in Nonhospitalized Patients. N Engl J Med. 2022 Feb 10;386(6):509-520. doi: 10.1056/NEJMoa2116044. Epub 2021 Dec 16. PMID 34914868
- [Background] Mahase E. Covid-19: Pfizer's paxlovid is 89% effective in patients at risk of serious illness, company reports. BMJ. 2021 Nov 8;375:n2713. doi: 10.1136/bmj.n2713. No abstract available. PMID 34750163
- [Background] Abbasi J. Studies Suggest COVID-19 Vaccine Boosters Save Lives. JAMA. 2022 Jan 11;327(2):115. doi: 10.1001/jama.2021.23455. No abstract available. PMID 35015054
- [Background] Burckhardt RM, Dennehy JJ, Poon LLM, Saif LJ, Enquist LW. Are COVID-19 Vaccine Boosters Needed? The Science behind Boosters. J Virol. 2022 Feb 9;96(3):e0197321. doi: 10.1128/JVI.01973-21. Epub 2021 Nov 24. PMID 34817198
- [Background] Mattiuzzi C, Lippi G. Efficacy of COVID-19 vaccine booster doses in older people. Eur Geriatr Med. 2022 Feb;13(1):275-278. doi: 10.1007/s41999-022-00615-7. Epub 2022 Jan 24. PMID 35067909
- [Background] Parker EPK, Desai S, Marti M, Nohynek H, Kaslow DC, Kochhar S, O'Brien KL, Hombach J, Wilder-Smith A. Response to additional COVID-19 vaccine doses in people who are immunocompromised: a rapid review. Lancet Glob Health. 2022 Mar;10(3):e326-e328. doi: 10.1016/S2214-109X(21)00593-3. No abstract available. PMID 35180408
- [Background] Fadlyana E, Rusmil K, Tarigan R, Rahmadi AR, Prodjosoewojo S, Sofiatin Y, Khrisna CV, Sari RM, Setyaningsih L, Surachman F, Bachtiar NS, Sukandar H, Megantara I, Murad C, Pangesti KNA, Setiawaty V, Sudigdoadi S, Hu Y, Gao Q, Kartasasmita CB. A phase III, observer-blind, randomized, placebo-controlled study of the efficacy, safety, and immunogenicity of SARS-CoV-2 inactivated vaccine in healthy adults aged 18-59 years: An interim analysis in Indonesia. Vaccine. 2021 Oct 22;39(44):6520-6528. doi: 10.1016/j.vaccine.2021.09.052. Epub 2021 Sep 24. PMID 34620531
- See also: New York Vaccine Tracker. Accessed 30 April 2022. — https://www.nytimes.com/interactive/2020/science/coronavirus-vaccine-tracker.html
- See also: Badan POM Republik Indonesia. Accessed 11 October 2021. — https://www.pom.go.id/siaran-pers/pastikan-keamanan-dan-mutu-vaksin-badan-pom-kawal-uji-klinik-vaksin-merah-putih
- See also: Worldometer coronavirus cases. Accessed 30 March 2023. — https://www.worldometers.info/coronavirus/
- See also: Our world in Data. Accessed 30 April 2022. — https://ourworldindata.org/covid-vaccinations
- See also: CNN. Accessed 11 October 2021. — https://edition.cnn.com/2021/04/03/health/us-coronavirus-saturday/index.html
- See also: World Health Organization. Accessed 11 October 2021. — https://www.who.int/news-room/feature-stories/detail/vaccine-efficacy-effectiveness-and-protection
- See also: Badan POM Republik Indonesia. Accessed 11 April 2022. — https://www.pom.go.id/siaran-pers/badan-pom-terbitkan-eua-vaksin-covovax-sebagai-vaksin-alternatif-ke-11-dalam-penanganan-pandemi
- See also: CNN Indonesia. Accessed 11 October 2021. — https://www.cnnindonesia.com/ekonomi/20210615172504-92-654688/bio-farma-yakin-ri-bisa-dapat-400-juta-dosis-vaksin-tahun-ini
- See also: Suara.com. Accessed 11 October 2021. — https://www.suara.com/bisnis/2020/11/06/151502/ini-6-lembaga-yang-kembangkan-vaksin-merah-putih